CLINICAL TRIAL: NCT04083027
Title: Patterns of Non-mass Enhancement of Breast MRI Using the BI-RADS Lexicon Fifth Edition With Histopathologic Correlation
Brief Title: Non-mass Enhancement in Breast MRI
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Gamal Hassan, Principal Investigator, Assiut University
Other Study IDs: Breast MRI
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: MRI — Breast MRI

SUMMARY:
Breast Magnetic Resonance Imaging (MRI) has been proven to be the most sensitive method in detection of breast cancer with sensitivity reaching 68-100%. The most frequent indication for breast MRI is screening for high-risk patients with a 20% or greater lifetime risk of developing breast cancer. Other indications include; assessment of extent of disease and screening of the contralateral breast in patients who are newly diagnosed with primary breast cancer. Evaluation of residual disease post Breast Conserving Surgery (BCS) with positive margins, loco-regional recurrence detection, as well as response to neoadjuvant chemotherapy are also well visualized by breast MRI. Furthermore, assessment of inconclusive mammography finding without a sonographic correlate, suspicious nipple discharge without a sono-mammographic or galacto-graphic correlate and evaluation of metastatic axillary lymphadenopathy in case of unknown primary tumor are all indications in which breast MRI has shown high sensitivity.

Breast MRI also helps in identifying multifocal/multicentric or contralateral breast malignancies which was not detected by conventional imaging. Moreover, MRI gives more accurate data about local extension of invasive breast cancer and in situ tumors than other conventional modalities. In some patients newly diagnosed to have cancer breast, breast MRI is able to detect additional lesions that has not been found in mammography or breast ultrasound in 6 - 34% in the ipsilateral breast and 3 - 5% in the contralateral breast. These additional breast lesions are classified into focus, mass, and non-mass enhancement (NME) on MRI.

Non-mass enhancement (NME) is defined as an enhancing abnormality that is not associated with the three-dimension volume of a mass, shape and outlining, and they are separate from the Background Parenchymal Enhancement (BPE). The fifth edition of the American College of Radiology (ACR) Breast Imaging-Reporting and Data System (BI-RADS) lexicon has erased some ambiguities, and modified terminologies from the fourth edition to provide more precise evaluation in descriptions of the distribution and Internal Enhancement Patterns (IEPs) of NME, contributes in quality assurance, better communication with physicians, and enhances patient care.

For morphological assessment of NME, distribution is described as focal, linear, segmental, regional, multiple regions, and diffuse. And the IEPs are characterized as homogeneous, heterogeneous, clumped, and clustered ring. NME may be benign as Pseudoangiomatous Stromal Hyperplasia (PASH), apocrine metaplasia and radiation effect; high risk such as Atypical Ductal Hyperplasia (ADH), flat epithelial atypia, intraductal papilloma, radial scar or complex sclerosing lesion, or malignant as Ductal Carcinoma in-situ (DCIS), Invasive Ductal Carcinoma (IDC), and Invasive Lobular Carcinoma (ILC).

ELIGIBILITY:
Inclusion Criteria:

* all female with mean age 50 ± 17 having breast MRI

Exclusion Criteria:

* Contraindications of MRI as pacemakers, aneurysmal clipping, retained metallic foreign bodies, or claustrophobic patients
* Pregnant women especially in the first trimester.

Ages: 33 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Female patients with mean age 50 ± 17
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Patterns of non-mass enhancement on breast MRI | Within one year; from March 2020 to March 2021
  To estimate the various patterns of NME using the BI-RADS lexicon fifth edition with histopathologic correlation; to evaluate their clinical significance.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park SY, Han BK, Ko ES, Ko EY, Cho EY. Additional lesions seen in magnetic resonance imaging of breast cancer patients: the role of second-look ultrasound and imaging-guided interventions. Ultrasonography. 2019 Jan;38(1):76-82. doi: 10.14366/usg.18002. Epub 2018 Jun 23. PMID 30103597
- [Background] Shin K, Phalak K, Hamame A, Whitman GJ. Interpretation of Breast MRI Utilizing the BI-RADS Fifth Edition Lexicon: How Are We Doing and Where Are We Headed? Curr Probl Diagn Radiol. 2017 Jan-Feb;46(1):26-34. doi: 10.1067/j.cpradiol.2015.12.001. Epub 2015 Dec 15. PMID 26826797
- [Background] Ha GW, Yi MS, Lee BK, Youn HJ, Jung SH. Clinical outcome of magnetic resonance imaging-detected additional lesions in breast cancer patients. J Breast Cancer. 2011 Sep;14(3):213-8. doi: 10.4048/jbc.2011.14.3.213. Epub 2011 Sep 29. PMID 22031803
- [Background] Cho YH, Cho KR, Park EK, Seo BK, Woo OH, Cho SB, Bae JW. Significance of Additional Non-Mass Enhancement in Patients with Breast Cancer on Preoperative 3T Dynamic Contrast Enhanced MRI of the Breast. Iran J Radiol. 2016 Jan 23;13(1):e30909. doi: 10.5812/iranjradiol.30909. eCollection 2016 Jan. PMID 27127579
- [Background] Lee SM, Nam KJ, Choo KS, Kim JY, Jeong DW, Kim HY, Kim JY. Patterns of malignant non-mass enhancement on 3-T breast MRI help predict invasiveness: using the BI-RADS lexicon fifth edition. Acta Radiol. 2018 Nov;59(11):1292-1299. doi: 10.1177/0284185118759139. Epub 2018 May 14. PMID 29758996
- [Background] Yang QX, Ji X, Feng LL, Zheng L, Zhou XQ, Wu Q, Chen X. Significant MRI indicators of malignancy for breast non-mass enhancement. J Xray Sci Technol. 2017;25(6):1033-1044. doi: 10.3233/XST-17311. PMID 29154312
- [Background] Machida Y, Shimauchi A, Tozaki M, Kuroki Y, Yoshida T, Fukuma E. Descriptors of Malignant Non-mass Enhancement of Breast MRI: Their Correlation to the Presence of Invasion. Acad Radiol. 2016 Jun;23(6):687-95. doi: 10.1016/j.acra.2016.01.014. Epub 2016 Mar 11. PMID 26976623
- [Background] D'Orsi CJ, Sickles EA, Mendelson EB, Morris EA, et al. ACR BI-RADS Atlas, Breast Imaging Reporting and Data System. Reston, VA, American College of Radiology; 2013.
- [Background] Chadashvili T, Ghosh E, Fein-Zachary V, Mehta TS, Venkataraman S, Dialani V, Slanetz PJ. Nonmass enhancement on breast MRI: review of patterns with radiologic-pathologic correlation and discussion of management. AJR Am J Roentgenol. 2015 Jan;204(1):219-27. doi: 10.2214/AJR.14.12656. PMID 25539260